CLINICAL TRIAL: NCT05827471
Title: Clinical Application of Sulfhydryl Oxidase QSOX1 as a New Biomarker of Colon Cancer
Brief Title: Clinical Study of QSOX1 as a Biomarker for Colon Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, YunqiuWang, Dr, Qianfoshan Hospital
Other Study IDs: QianfoshanHwyq20230305
Record Dates: First submitted 2023-03-26; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples and colon tissue samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tumor group: First diagnosis of colon cancer.
  Interventions: Diagnostic Test: Diagnosis of colon cancer
- Control group: Healthy people.
  Interventions: Diagnostic Test: Diagnosis of colon cancer

INTERVENTIONS:
Diagnostic Test: Diagnosis of colon cancer — Clinical diagnosis results

SUMMARY:
The goal of this observational study is to determine whether the secreted protein QSOX1 can be used as a molecular marker for early rapid diagnosis and accurate treatment of colon cancer.

DETAILED DESCRIPTION:
The project mainly selects the tumor group represented by colon cancer and the corresponding healthy people as the control group, with about 100 cases in each of the two groups. Mainly collect blood and tumor tissue samples of patients, detect the expression of QSOX1 in the above samples, and explore the role in the diagnosis and prognosis evaluation of colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* Colon cancer was confirmed by colonoscopic pathology.
* No local or systemic treatment was performed before operation.
* Complete clinical data.

Exclusion Criteria:

* Combined with benign diseases of colon, such as ulcerative colitis, colon adenoma and colon polyp.
* Other tumors other than colon cancer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients diagnosed with colon cancer for the first time admitted to the First Affiliated Hospital of Shandong First Medical University.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of RNA for early rapid diagnosis of colon cancer. | 6 months
  RT-PCR was used to detect the RNA levels of QSOX1 in the tumor and control groups.
Detection of protein for early rapid diagnosis of colon cancer. | 6 months
  Western blotting was used to detect the protein levels of QSOX1 in the tumor and control groups.